CLINICAL TRIAL: NCT05316090
Title: Effect of Core Stability Excercises Program on Reaching in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Lecturer of pediatric physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003125
Record Dates: First submitted 2022-03-23; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: study group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Children in study group treated using core stability exercises program in addition to traditional program
  Interventions: Procedure: Core stability exercises program; Procedure: Traditional physical therapy program
- control group (Active Comparator): Children in the control group treated using traditional physical therapy program.
  Interventions: Procedure: Traditional physical therapy program

INTERVENTIONS:
Procedure: Core stability exercises program — Strengthening to the trunk muscles
  Arms: study group
Procedure: Traditional physical therapy program — Neurodevelopmental training excercises

SUMMARY:
Purpose of the study:

To evaluate effect of core stability exercises program on upper limb reaching in children with spastic hemiparetic cerebral palsy.

DETAILED DESCRIPTION:
Thirty spastic hemiparetic cerebral palsied children of both sexes will be selected from General hospitals and private centers in El-Minia government with the following criteria:

1. The age of the selected children ranged from 3 To 6 years old.
2. Degree of spasticity is ranging from 1 to 1+, according to modified Ashworth scale
3. Children in study group will be treated using core stability exercises program in addition to traditional program and children in the control group will be treated using traditional physical therapy program.
4. Trunk control measurement scale and pediatric reach test will be used to evaluate each child individually before and after 6 successive weeks of treatment, three times per week.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the selected children ranged from 3 To 6 years old.
2. Degree of spasticity is ranging from 1 to 1+, according to modified Ashworth scale(Bohannon and Smith, 1987).
3. Children with hemiparetic cerebral palsy

Exclusion Criteria:

1. Fructures and fixed deformities

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-08 (Actual)

PRIMARY OUTCOMES:
Pediatric reach test | assessment after 6 weeks of intervention
  Reaching score

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abbass, Ph.D., Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No